CLINICAL TRIAL: NCT06043739
Title: A Randomized, Open-label, 3-period, Single-dose, Cross-over Study in Healthy Adult Subjects to Assess the Relative Bioavailability of Filgotinib Given as an Oral Mini-tablet Formulation Versus the Oral Tablet Formulation of Filgotinib and to Assess the Effect of Food on the Oral Mini-tablet Formulation
Brief Title: Relative Bioavailability and Effect of Food Study With an Oral Mini-tablet Formulation of Filgotinib in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GLPG0634-CL-124
Record Dates: First submitted 2023-09-11; First posted 2023-09-21 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Bioavailability
MeSH Terms: interventions — GLPG0634

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment A: (Active Comparator): filgotinib administered under fasting conditions
  Interventions: Drug: Filgotinib
- Treatment B: (Experimental): filgotinib administered under fasting conditions
  Interventions: Drug: Filgotinib
- Treatment C: (Experimental): filgotinib administered under high-fat fed conditions
  Interventions: Drug: Filgotinib

INTERVENTIONS:
Drug: Filgotinib — Commercially developed film-coated tablet administered orally
  Other Names: GS-6034; GLPG0634; Jyseleca
  Arms: Treatment A:
Drug: Filgotinib — Film-coated mini-tablets administered orally
  Other Names: GS-6034; GLPG0634
  Arms: Treatment B:; Treatment C:

SUMMARY:
Open label study to assess relative bioavailability of filgotinib oral mini-tablet versus oral tablet formulation and effect of food on the mini-tablet formulation.

ELIGIBILITY:
Key Inclusion Criteria:

* A body mass index (BMI) between 18.0 and 30.0 kg/m2, inclusive.
* Judged to be in good health by the investigator based upon the results of a medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG), and fasting clinical laboratory safety tests. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) must be no greater than 1.5x upper limit of normal range (ULN) and total bilirubin not greater than ULN. Other clinical laboratory safety test results must be within the normal ranges or test results that are outside the normal ranges need to be considered not clinically significant in the opinion of the investigator.

Key Exclusion Criteria:

* Known hypersensitivity to filgotinib ingredients or history of a significant allergic reaction to filgotinib ingredients as determined by the investigator.
* Treatment with any medication (including over-the-counter (OTC) and/or prescription medication, dietary supplements, nutraceuticals, vitamins and/or herbal supplements) except occasional paracetamol (maximum dose of 2 g/day and maximum of 10 g/2 weeks) in the last 2 weeks or 5 half-lives of the drug, whichever is longer, prior to the first dosing.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-09-22 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2023-11-12 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration of filgotinib (Cmax) | From Day 1 pre-dose until Day 15
Cmax of GS-829845, major active metabolite | From Day 1 pre-dose until Day 15
Area under the plasma concentration-time curve from time zero till the last observed quantifiable concentration of filgotinib (AUC0-t) | From Day 1 pre-dose until Day 15
AUC0-t of GS-829845, major active metabolite | From Day 1 pre-dose until Day 15
Area under the plasma concentration time curve from time zero to infinity of filgotinib (AUC0-inf) | From Day 1 pre-dose until Day 15
AUC0-inf of GS-829845, major active metabolite | From Day 1 pre-dose until Day 15

SECONDARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs), treatment-emergent serious adverse events (SAEs), and TEAEs leading to treatment discontinuations | Baseline (Day 1) up to 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Galapagos Study Director, Study Director — Galapagos NV
Locations (1):
- Altasciences, Montreal, Canada

IPD SHARING:
Plan to Share IPD: No